CLINICAL TRIAL: NCT04570189
Title: Evaluating Auscul-X, a Touch Free Digital Stethoscope, for Physical Distancing to Protect Patients and Health Care Professionals From COVID-19 (The Auscul-X Study)
Brief Title: Evaluating Auscul-X, a Touch Free Digital Stethoscope
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AusculSciences Canada Inc. (Industry)
Collaborators: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Sponsor
Other Study IDs: Auscul-X
Record Dates: First submitted 2020-09-17; First posted 2020-09-30 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Phase I: Twenty subjects, 10 unventilated and 10 ventilated patients, will undergo clinical auscultation of the heart and lungs with the Auscul-X, a conventional stethoscope and an electronic stethoscope (Littmann 3200).
  Interventions: Device: Auscul-X
- Phase II: Twenty subjects, 10 unventilated and 10 ventilated patients, will undergo clinical auscultation of the heart and lungs with an Auscul-X with wireless capability, a conventional stethoscope and an electronic stethoscope (Littmann 3200). Phase II shall begin upon appropriate Health Canada approvals for the Auscul-X with wireless capability.
  Interventions: Device: Auscul-X

INTERVENTIONS:
Device: Auscul-X — The Auscul-X System (AusculSciences Canada, Inc.), is novel, professional grade, touch free, multichannel, touch-free electronic stethoscope with disposable elements designed to protect HCPs from exposure to infection diseases by allowing them to auscultate patients from a safe distance (10 feet away). The sensors can stay in place and enable providers to listen on-demand to a patient's heart and lungs over an extended period of time. This practice of distancing in the workplace is a key CDC and PHAC recommendation to protect the frontline HCP from exposure risk to the highly contagious COVID- 19 virus and other communicable diseases. The Auscul-X not only has the potential to better protect HCPs from infection, but also eliminates the potential transmission of pathogens through the use of conventional stethoscopes. In addition, the Auscul-X allows multiple HCPs to listen to the patient's heart and lung sounds simultaneously

SUMMARY:
Auscul-X a touch free digital stethoscope will permit physical distancing of healthcare providers while maintaining the ability to auscultate patients from a safe distance (over 10 feet away)

DETAILED DESCRIPTION:
The Auscul-X System (AusculSciences Canada, Inc.), is novel, professional grade, touch free, multichannel, touch-free electronic stethoscope with disposable elements designed to protect HCPs from exposure to infection diseases by allowing them to auscultate patients from a safe distance (10 feet away). The sensors can stay in place and enable providers to listen on-demand to a patient's heart and lungs over an extended period of time. This practice of distancing in the workplace is a key CDC and PHAC recommendation to protect the frontline HCP from exposure risk to the highly contagious COVID- 19 virus and other communicable diseases. The Auscul-X not only has the potential to better protect HCPs from infection, but also eliminates the potential transmission of pathogens through the use of conventional stethoscopes. In addition, the Auscul-X allows multiple HCPs to listen to the patient's heart and lung sounds simultaneously

ELIGIBILITY:
Inclusion Criteria:

* >/=18 years old
* Admitted to ICCU and CSICU at UOHI

Exclusion Criteria:

* Age < 18 years old
* Medically Unstable
* Chest wall deformity or wounds in adhesive application areas
* Unwillingness or inability to provide Informed Consent or to comply with protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study will recruit 40 (Phase 1 = 20 patients, Phase 2 = 20 patients) adult participants age 18 years old, who are under care in the Intensive Cardiac Care Unit (ICCU) or Cardiac Surgical Intensive Care Unit (CSICU) at the University of Ottawa Heart Institute.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility and use of Auscul-X for listening to heart and lung sounds will be assessed by ICU clinicians to determine Auscul-X is at least equivalent to a digital stethoscope using a Likert scale for comparison. | up to 1 Year
  To determine the feasibility of implementing Auscul-X in the critical/intensive care environment (ICCU and CSICU).

SECONDARY OUTCOMES:
The measurement for acoustic quality in high risk settings determined as clarity and loudness by means of a Likert scale for comparison of Auscul-X and digital stethoscopes by clinicians. | up to 1 year
  1. Determine if the quality of the real-time heart and lung sounds (Likert scale) for the Auscul-X will be similar to the conventional stethoscope and digital electronic stethoscope in the ICCU and CSICU (Appendix A).
  2. Determine if the acoustic recordings taken as part of Phase II for the Auscul-X and conventional electronic stethoscope are similar (as evaluated by independent blinded cardiologists and respirologists using a Likert scale for acoustic and diagnostic quality (Appendix B)).
  3. Determine if the acoustic recordings for the Auscul-X and conventional electronic stethoscope provide similar signal quality using objective acoustic metrics (e.g. signal to noise ratios, etc.) (Phase II only)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Chow, MD, Principal Investigator — Ottawa Heart Institue Research Foundation
Locations (1):
- The University of Ottawa Heart Institute, Ottawa, Ontario, Canada